CLINICAL TRIAL: NCT05480618
Title: Effect of Slow Breathing and Yogic-Derived Breathing on Respiration and Cardiovascular Variability in Spinal Cord Injury Patients
Brief Title: Slow Yogic-Derived Breathing and Respiration and Cardiovascular Variability in Spinal Cord Injury Patients
Acronym: SCOGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, J. Andrew Taylor, Associate Professor of Physical Medicine and Rehabilitation, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022P001696
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries; Slow Breathing
Keywords: resonance; yogic; pranayama; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Hypoventilation

STUDY DESIGN:
Intervention Model Description: This study will be a small prospective cohort (N= 20) study with a one-time unblinded intervention of 4 differing breathing techniques/ratios compared to spontaneous breathing. Patients will receive instruction on D1 and on D7 lasting about 45 minutes and a diary for self-practice. On D14 the participant will be asked to sequentially perform the directed breathing frequencies and ratios. The lab visit will last approximately 1.5 hours, during which beat-by-beat cardiovascular variables and breath-by-breath respiratory variables will be recorded. The total in-person time commitment (~4 hours) over the 14 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal Cord Injury Subjects (Experimental): 20 medically stable male and female subjects between 18 and 60 years old, BMI between 18.5-35 kg/m2, with a history of SCI and who use a wheelchair were included. Participants that did not speak English or with a history of renal, neurological, or coronary artery disease, cancer, diabetes, significant arrhythmia smoking, or using cardioactive medications were excluded.
  Interventions: Behavioral: Slow Breathing

INTERVENTIONS:
Behavioral: Slow Breathing — On two separate visits (on Day 1 and between Day 7 and 9 of their self-practice) the subject will be coached on yoga breathing techniques.
  The breathing techniques will be varied in:
  1. frequency (between 0.25 and 0.1 Hz)
  2. Inspiratory:Expiratory (I:E) ratio or 'Duty Cycle'
  3. with and without ujjayi (yogic throat restriction)
  4. with and without inspiratory/expiratory breath holding
  At the end of the first coaching visit the subject will be given a diary to record their own practice of the breathing techniques they were coached on.
  Other Names: Yogic-Derived Breathing

SUMMARY:
This research will aid in understanding of slow-breathing and its effect on heart rate and blood pressure in people with a spinal cord injury (SCI). This research will investigate if traditional 'yogic' breathing exercises can be performed by subjects with SCI and its influence on the cardiovascular system.

DETAILED DESCRIPTION:
The relationship between respiratory patterns and cardiovascular variability in healthy persons has been previously studied. However, the impact of SCI on the interrelationships between the respiratory and cardiovascular systems remains relatively unstudied. The loss of autonomic control in SCI may mean that slow breathing has profound effects on cardiovascular variability. Hence, those with SCI may represent a population that could benefit from the potential physiologic effects of numerous yogic-based breathing patterns that can be applied anywhere any time. Hence, it is important to determine if slower breathing patterns can shift the cardiovascular control pattern to-wards important healthful effects. This physiological study will compare the effects of uncontrolled breathing and traditional yogic slow-breathing practices on cardiovascular variability in SCI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years old
2. Wheelchair user
3. Medically stable & able to follow directions
4. Body mass index (18.5 - 35 kg/m2)

Exclusion Criteria:

1. BP >140/90 mmHg
2. Current use of cardioactive medications (except medication to support blood pressure)
3. Current tobacco use
4. Significant arrhythmia
5. Coronary artery disease
6. Diabetes
7. Renal Disease
8. Cancer
9. Epilepsy or other neurological diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | 1,5 hour during Slow-breathing
  R-R interval on a 5 lead Electrocardiogram (EKG)
beat-by-beat arterial pressure | 1,5 hour during Slow-breathing
  blood pressure fluctuations via Finometer and Dinamap blood pressure cuff
beat-by-beat limb blood flow | 1,5 hour during Slow-breathing
  brachial blood flow via doppler
peripheral capillary oxygen saturation (SpO2) | 1,5 hour during Slow-breathing
  blood oxygen saturation via pulse oximetry
respiratory excursions | 1,5 hour during Slow-breathing
  Measuring belly and chest depth of inspiration and expiration

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazur MD, Hamner JW, Anand AN, Taylor JA. Cardiorespiratory Effects of Yogic Versus Slow Breathing in Individuals with a Spinal Cord Injury: An Exploratory Cohort Study. J Integr Complement Med. 2024 Sep;30(9):878-885. doi: 10.1089/jicm.2023.0641. Epub 2024 Mar 20. PMID 38507692